CLINICAL TRIAL: NCT06820164
Title: Lipomas Treated with Subcutaneous Injections of Cooled Sodium Chloride: an Exploratory Study
Brief Title: Lipomas Treated with Subcutaneous Injections of Cooled Sodium Chloride
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Jessica Patterson, Assistant Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2410045096
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Lipoma
MeSH Terms: conditions — Lipoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cooled Sodium Chloride Injection (Experimental): Injection of a solution containing sterile, cooled 0.9% sodium chloride and 1% lidocaine with epinephrine (1:100,000). Each patient will receive a volume of solution equal to three times the estimated volume of the lipoma; the first cc of the injection will be lidocaine with epinephrine, and the remainder will be sterile normal saline. The solution will be cooled using an ice/saline bath at -1°C. Following the injection, the lipoma will be gently massaged for one minute to distribute the saline evenly.
  Interventions: Drug: Cooled Sodium Chloride Injection

INTERVENTIONS:
Drug: Cooled Sodium Chloride Injection — Injection of a solution containing sterile, cooled 0.9% sodium chloride and 1% lidocaine with epinephrine (1:100,000).

SUMMARY:
Lipomas are benign tumors composed of mature adipose tissue. While harmless, these are the most common type of soft tissue growths with some patients developing numerous lipomas. Patients often seek removal for cosmesis, or symptoms caused by location and/or compression of surrounding structures. This exploratory study aims to evaluate the effectiveness of subcutaneous injections of cooled normal saline as a treatment option for lipomas. The study will assess whether this technique could serve as a viable alternative to existing treatment options, especially compared to topically applied fat-freezing devices. The Investigators propose that this method may offer a more comfortable nonsurgical option for targeted fat reduction, as the cold temperatures are applied directly to the lipomas.

ELIGIBILITY:
Inclusion Criteria:

* At least one clinically diagnosed subcutaneous lipoma

Exclusion Criteria:

* Unable to give informed consent
* Participant has a lipoma on the face
* Lipomas located subfascial or within deep tissue (e.g., intramuscular lipomas)
* Lipomas larger than 10 cm in diameter (fat deposits exceeding 500 mL in volume)
* Rapidly growing lipomas
* Lipomas exhibiting abnormal ultrasound findings (e.g., complex hyperechoic patterns, internal heterogeneity, or multilobulated appearance)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Post-Injection Pain (First Treatment) | 15 minutes post injection (treatment)
  Pain is assessed using a scale of 0-10 reported by the patient, with 0 being no pain and 10 being the worst pain ever experienced.
Post-Injection Pain (Second Treatment) | 15 minutes post injection (treatment)
  Pain is assessed using a scale of 0-10 reported by the patient, with 0 being no pain and 10 being the worst pain ever experienced.
Post-Injection Pain (Third Treatment) | 15 minutes post injection (treatment)
  Pain is assessed using a scale of 0-10 reported by the patient, with 0 being no pain and 10 being the worst pain ever experienced.
Post-injection erythema (First Treatment) | 15 minutes post injection (treatment)
  Post-injection erythema is assessed using a scale of 0-4 as per the Clinical Erythema Assessment grading scale with: 0 = clear, 1 = almost clear, 2 = mild erythema, 3 = moderate erythema, and 4 = severe erythema. The higher score indicates a worse outcome.
Post-injection erythema (Second Treatment) | 15 minutes post injection (treatment)
  Post-injection erythema is assessed using a scale of 0-4 as per the Clinical Erythema Assessment grading scale with: 0 = clear, 1 = almost clear, 2 = mild erythema, 3 = moderate erythema, and 4 = severe erythema. The higher score indicates a worse outcome.
Post-injection erythema (Third Treatment) | 15 minutes post injection (treatment)
  Post-injection erythema is assessed using a scale of 0-4 as per the Clinical Erythema Assessment grading scale with: 0 = clear, 1 = almost clear, 2 = mild erythema, 3 = moderate erythema, and 4 = severe erythema. The higher score indicates a worse outcome.
Change in Lipoma Size | Baseline to Second Treatment (4-week interval between treatments)
  Change in Lipoma Size from the First Treatment (Baseline) to the Second Treatment. There is a 4 week interval between each treatment. Lipoma size is assessed using approximate lipoma area (cm × cm) determined by ultrasound, with the final percentage change being the following quotient: [(final area - initial area) ÷ initial area] × 100.
Change in Lipoma Size | Baseline to Third Treatment (4-week interval between treatments)
  Change in Lipoma Size from the First Treatment (Baseline) to the Third Treatment. Lipoma size is assessed using approximate lipoma area (cm × cm) determined by ultrasound, with the final percentage change being the following quotient: [(final area - initial area) ÷ initial area] × 100.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Patterson, MD, Principal Investigator — West Virginia University-Dermatology
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No